CLINICAL TRIAL: NCT01894763
Title: Randomized, Prospective Comparison of Large vs. Small Diameter Esophageal Stents for Palliation of Malignant Dysphagia
Brief Title: Prospective Comparison of Large vs. Small Diameter Esophageal Stents for Palliation of Malignant Dysphagia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Tenwek Hospital, Bomet, Kenya (Unknown)
Responsible Party: Principal Investigator, Mark Topazian, Professor of Medicine, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1063-04
Record Dates: First submitted 2013-06-26; First posted 2013-07-10 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2013-07

CONDITIONS: Esophageal Cancer
Keywords: esophagus; cancer
MeSH Terms: conditions — Esophageal Neoplasms; Neoplasms | interventions — Self Expandable Metallic Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Small-diameter stent (Active Comparator): Placement of a 23 mm self-expandable metal stent
  Interventions: Device: Self-expandable metal stent
- Large-diameter stent (Active Comparator): Placement of a 28-mm self-expandable metal stent
  Interventions: Device: Self-expandable metal stent

INTERVENTIONS:
Device: Self-expandable metal stent — Placement of a self-expandable metal stent in the esophagus
  Other Names: Ultraflex Esophageal Stents

SUMMARY:
Esophageal cancer often causes difficulty swallowing (dysphagia) that can be relieved by placement of a stent (a flexible, expandable tube that props open the blockage caused by the cancer). Stents are effective but can cause complications. Stents come in different diameters. The purpose of this study is to learn if stents of different diameters are more or less effective for treatment of dysphagia caused by esophageal cancer.

DETAILED DESCRIPTION:
This prospective, randomized study was conducted at Tenwek Hospital in Bomet, Kenya, and was approved by the hospital's institutional review board (IRB) as well as the Kenya Medical Research Institute's Ethical Review Committee. Participants with dysphagia were recruited and provided signed informed consent prior to endoscopy. During endoscopy and after dilation of an obstructing esophageal tumor sufficient to permit passage of an endoscope, eligible participants were enrolled and randomized to receive either an 18 mm shaft/23 mm flange or 23 mm shaft/28 mm flange partially covered Ultraflex esophageal stent (Boston Scientific, Natick, Massachusets, USA). Stents were either 10 or 12 cm in length, and the endoscopist chose a stent length based on the length of the malignant stricture. One stent was placed in each subject. Follow-up was then obtained at scheduled intervals after stent placement (7 and 28 days, 3 months, then every 3 months), until the participant's death. Earlier follow-up visits were arranged if participants reported any new health concerns.

Block randomization was performed using the sealed envelope technique, with 10 participants in each block; none of the study personnel at Tenwek Hospital had knowledge of the randomization sequence. Allocation was concealed from participants, caregivers, and study personnel until randomization occurred during an endoscopic procedure. After randomization, stent diameters were known to the endoscopy staff and listed in the medical record. All randomized participants correctly received a stent of the allocated diameter, and remained blinded to the stent diameter they received.

At baseline and each follow-up visit body weight was recorded, as well as Karnofsky performance status score, dysphagia score (0=normal, no dysphagia; 1=can swallow most foods; 2=can swallow a soft diet; 3=can swallow fluids only; 4=unable to swallow saliva), current medications, and the presence or absence of 15 symptoms and 9 diagnoses (weakness, fever, vomiting, vomiting blood, melena, weak voice, difficulty breathing, cough, sputum, palpitations, heartburn, chest pain, hiccoughs, recurrent dysphagia, abdominal pain; anemia, gastrointestinal bleeding, esophago-respiratory fistula, arrhythmia, pneumonia, metastases, stent occlusion, stent migration, gastroesophageal reflux disease). In addition, all interval clinic visits, test results, endoscopy reports, and hospitalizations were reviewed.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* dysphagia due to unresectable esophageal cancer
* participant resides within 50 km of Tenwek Hospital
* tumor is ≤ 9 cm in length and > 2 cm distal to the upper esophageal sphincter (UES)
* no esophago-respiratory fistula (ERF) or suspected perforation is present

Exclusion Criteria:

* unable to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2003-09; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Relief of dysphagia | 1 month following stent placement
  Number of participants with improvement in dysphagia score to <2
Complications | from stent placement to death or 5 years of follow-up, whichever comes first
  Number of participants who experience stent-related symptoms (including chest pain, recurrent dysphagia, hematemesis, melena, palpitations) or complications (including gastrointestinal hemorrhage, esophago-respiratory fistula, stent migration, stent occlusion) from the time of stent placement until death or 5-year follow-up.
Mortality | from stent placement to death or 5 years of follow-up, whichever comes first
  Time (in days) from stent placement to death, assessed by Kaplan-Meier analysis

SECONDARY OUTCOMES:
Endoscopic re-intervention | from stent placement to death or 5 years of follow-up, whichever comes first
  Number of participants undergoing repeat endoscopy to diagnose or treat a stent-related problem at any time from stent placement to death or 5 year follow-up.
performance status | from stent placement to death or 5 years of follow-up, whichever comes first
  Karnofsky performance status, assessed by Kaplan Meier analysis, from stent placement to death or 5-year follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Russell White, M.D., Principal Investigator — Tenwek Hospital, Bomet, Kenya
Locations (1):
- Tenwek Hospital, Bomet, Kenya

REFERENCES:
- [Derived] White RE, Chepkwony R, Mwachiro M, Burgert SL, Enders FT, Topazian M. Randomized Trial of Small-diameter Versus Large-diameter Esophageal Stents for Palliation of Malignant Esophageal Obstruction. J Clin Gastroenterol. 2015 Sep;49(8):660-5. doi: 10.1097/MCG.0000000000000333. PMID 25992812